CLINICAL TRIAL: NCT03121066
Title: Intervention Based on Transcranial Magnetic Stimulation for Alzheimer's Disease Patients: Randomized Clinical Trial
Brief Title: Transcranial Magnetic Stimulation for Alzheimer's Disease Treatment
Acronym: TMSAD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Universitat Oberta de Catalunya (Other)
Collaborators: Consorci Sanitari de Terrassa (Other)
Responsible Party: Principal Investigator, Elena Munoz Marron, Principal Investigator, Universitat Oberta de Catalunya
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UOCatalunya
Record Dates: First submitted 2017-04-01; First posted 2017-04-19 (Actual); Last update posted 2022-11-09 (Actual); Status verified 2022-11

CONDITIONS: Alzheimer Disease
Keywords: Transcranial Magnetic Stimulation; Non invasive brain stimulation; Theta Burst Protocol; Brain connectivity; Dorsolateral prefrontal cortex; Parietal cortex
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Intervention Model Description: The design of the study is a randomized, double blind, parallel clinical trial.
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Experimental group (Active Comparator): Transcranial Magnetic Stimulation + Conventional intervention
  Interventions: Device: Active Transcranial Magnetic Stimulation
- Sham control group (Sham Comparator): Sham Transcranial Magnetic Stimulation + Conventional intervention
  Interventions: Device: Sham Transcranial Magnetic Stimulation
- Non TMS Control group (No Intervention): Conventional intervention alone

INTERVENTIONS:
Device: Active Transcranial Magnetic Stimulation — The intervention consists of a 2-week treatment during which TMS will be applied for 10 days (every working day). The stimulation protocol will be intermittent TBS (iTBS). 600 pulses in each area will be applied at intervals of 2 seconds of stimulation and 8 seconds of rest; the total number of pulses per session will be 1200. The stimulation duration is 3 minutes and 12 seconds. This protocol allows the induction of long-term potentiation effects, promoting plasticity in the stimulated areas. To perform the stimulation a 70 mm, figure of 8-coil will be used. In order to precisely locate the stimulated areas a stereotactic image guidance will be used during the stimulation (Brainsight™ 2)
  Other Names: Magstim Super Rapid 2
  Arms: Experimental group
Device: Sham Transcranial Magnetic Stimulation — The Sham intervention will be carried out using the same stimulation protocol as in the active condition but with the coil rotated 90º to prevent the magnetic field inducing electrical activity in the cortex.
  Other Names: Magstim Super Rapid 2
  Arms: Sham control group

SUMMARY:
Background: Alzheimer's disease is a major health problem in our society. To date, pharmacological treatments to reduce Alzheimer's disease symptoms have obtained poor results and there is a growing interest in finding non-pharmacological treatments for this impactful disease. Transcranial Magnetic Stimulation is a non-invasive tool which can induce changes in brain activity and long term modifications of impaired neural networks, and therefore holds promise as a clinical intervention.

Our overall goal is to study the benefit of targeting Transcranial Magnetic Stimulation based on the individual's unique functional connectivity (personalized targeting) instead of current non-individualized approaches. Specifically, the intermittent Theta Burst protocol will be used and changes in cognitive, functional, and emotional deficits in these patients will be evaluated. Functional brain connectivity changes induced by the TMS treatment will be also assessed.

Methods: A double blind randomized controlled trial will be conducted to assess the effects of TMS treatment immediately, one month, three months and six months after the end of the treatment in comparison to the baseline measurements. Forty-five patients with a diagnosis of Alzheimer's disease, will be randomly allocated (1:1:1) into experimental (active Transcranial Magnetic Stimulation), sham control group, or conventional intervention control group. Neuropsychological, functional, and emotional assessment will be conducted, as well as functional connectivity measures, in order to assess the effectiveness of the treatment.

Discussion: The investigators expect to demonstrate that personalized Transcranial Magnetic Stimulation intervention has measurable positive impact in cognitive and emotional functioning, functionality, and brain connectivity, thus representing a potential treatment for Alzheimer's disease.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Alzheimer's disease according to the diagnostic criteria of the National Institute on Ageing and the Alzheimer's Association
* Ages between 60 and 75 years
* Mini Mental State Examination score between 20 and 26
* Global Deterioration Scale score of 3 or 4
* Functional independence for basic daily life activities (part C of the Blessed Scale equal or 0)
* Rosen Ischemia Scale less or equal to 4
* Able to read and write
* Stable medical and pharmacological state during the 3 consecutive months immediately before the start of the study
* Computed Tomography Scan and Magnetic Resonance Imaging in the last 12 months previous to the selection, compatible with the diagnosis of probable Alzheimer's disease in the subjects diagnosed
* Absence of clinically significant anomalies in the medical history or clinical laboratory results during the selection
* Screening analyses within normal range with the objective of detecting and excluding other causes of dementia in the last 12 months previous to selection. Laboratory values required in order to be considered within the normal range are as follows: complete blood count, thyroid hormones, T4, folic acid, vitamin B12, albumin, transaminase alanine, amino-transferase aspartate, gamma-glutamic transferase, sodium, potassium, urea, creatinine, glucose while fasting
* Being treated by Acetylcholinesterase Inhibitors
* Signed consent form, previously approved by the Research Ethics Committee

Exclusion Criteria:

* Knowledge of Spanish or Catalan after the age of 15
* Less than 4 years of schooling
* Intellectual deficiency (Premorbid Intelligence Quotient, vocabulary, less than 85)
* Not controlled medical conditions or severe mental disorders that may affect the Central Nervous System, including signs of increased intracranial pressure or intracranial lesions
* Presenting one or more vascular risks
* Medical conditions not controlled that may cause medical emergencies in case the produce convulsions (expel: cardiac malformations, cardiac arrhythmias, asthma, etc.)
* Medical history of convulsions, previous diagnosis of epilepsy, previous registry of abnormal electroencephalogram or family history of epilepsy
* Severe hearing problems or ringing in the ears (tinnitus)
* Severe loss of visual acuity
* Moderate or severe depression according to a score >11 (moderate depression) or 19 (severe depression) in the Geriatric Depression Scale
* Presence of tremors or motor control of the dominant upper extremity
* Being under pharmacological treatment with medications indicated in the security guidelines.
* Drug or alcohol consumption or history of abuse in the last 24 months prior to the study
* Implants of metal pieces in the brain (excluding dental fillings)
* Either of the following medical devices: pacemaker, implanted medication pumps, vagal nerve stimulators, deep cerebral stimulators, transcutaneous electrical stimulation units, ventriculus-peritoneal derivations, titanium plates, cochlear implants, aneurysm clips, etc…
* Negative response towards new technology
* Existence of any situation that may cause the subject, according to the principal researcher, not be an adequate candidate for the study

Ages: 60 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2023-11 (Estimated); Primary Completion 2024-09 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Change in Cognitive improvement | Baseline and 1 month, 3 months and 6 months after the end of the treatment
  Changes in cognitive functions will be assessed through a Neuropsychological Batery

SECONDARY OUTCOMES:
Functional capacity changes_1 | Baseline and 1 month, 3 months and 6 months after the end of the treatment
  Functional capacity will be assessed through the Functional Assessment Questionnaire (FAQ)
Functional capacity changes_2 | Baseline and 1 month, 3 months and 6 months after the end of the treatment
  Functional capacity will be assessed through the UCSD Performance-Based Skills Assessment (UPSA)
Mood changes | Baseline and 1 month, 3 months and 6 months after the end of the treatment
  Mood changes will be assessed through the Hospital Anxiety and Depression Scale (HAD)
Changes in brain connectivity | 3 days after the end of the treatment
  Brain connectivity will be assessed through the registry of brain activity in the resting state Magnetic Resonance Imaging.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Marron EM, Viejo-Sobera R, Quintana M, Redolar-Ripoll D, Rodriguez D, Garolera M. Transcranial magnetic stimulation intervention in Alzheimer's disease: a research proposal for a randomized controlled trial. BMC Res Notes. 2018 Sep 5;11(1):648. doi: 10.1186/s13104-018-3757-z. PMID 30185210